CLINICAL TRIAL: NCT00692029
Title: Kinematics of Youth (Age 12-15) on Stationary All Terrain Vehicles
Acronym: ATV
Status: Completed | Type: Observational
Sponsor: University of Kentucky (Other)
Responsible Party: Andrew Bernard, M.D., University of Kentucky
Other Study IDs: 08-0300-F1V
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-02

CONDITIONS: Healthy
Keywords: Normal; Healthy Volunteers

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
To assess the relationship between pre-teen/teen height, age, weight, gender, and body proportions and shape and size of youth and comfort and safety when operating adult All Terrain Vehicles (ATV).

ELIGIBILITY:
Inclusion Criteria:

1. males
2. age 12-15
3. a minimum level of physical skill to mount and dismount the vehicle
4. ability to speak and understand English.

We have used this age group because it is the most often injured group and represents an entire age group for ATV size restriction (other age groups not studied here are 6-11, and 16 or greater).

Exclusion Criteria:

1. inability to participate in physical education without restrictions
2. visual acuity < 20/40 corrected
3. females
4. emancipated minors.

We have excluded females to gain the most consistent body dimensions in this preliminary study.

Ages: 12 Years to 15 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Study Population: PreTeen and Teenage children
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2008-06; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
Quantify relationship of youth size/shape to comfort and safety when operating adult ATV | 1 session

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C. Bernard, M.D., Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States